CLINICAL TRIAL: NCT03232047
Title: A Randomized Control Trial on Computerized Cognitive Training for Individuals With Mild Cognitive Impairment
Brief Title: Computerized Cognitive Training for MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Huali Wang, Director of Clinical Research Division, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Z161100000516001
Record Dates: First submitted 2017-07-22; First posted 2017-07-27 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Computerized, Executive function, memory, cognitive training; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined cognitive training (Experimental): The training is combined executive function and memory training. The training is considered 'adaptive', which means that the difficulty level of the tasks increases during the sessions according to the individual level of mastering for each participant, making the patient work at their maximum capacity at all times.
  Interventions: Device: Combined executive function and memory training
- Waiting-list group (No Intervention): Participants in the control condition will conduct the same training as the intervention group after a 26-week waiting period. During the 26-week waiting period, the participants will receive assessment with the same protocol as the interventional group.

INTERVENTIONS:
Device: Combined executive function and memory training — Computerized combined executive function and memory training
  Arms: Combined cognitive training

SUMMARY:
The objective of the study is to evaluate whether memory training combined with executive training could lead to improved cognitive and noncognitive performance in patients with MCI. Furthermore, we will explore the neural correlates underlying the changed performances.

DETAILED DESCRIPTION:
Introduction:

Mild cognitive impairment (MCI) is a clinical condition characterized of a reduction in memory and/or other cognitive processes that are insufficiently severe to be diagnosed as dementia, but are more pronounced than the cognitive decline associated with normal aging. The prevalence of MCI ranges from 3% to 19% in adults older than 65 years; some of these individuals seem to remain stable or return to normal over time, but more than half progress to dementia within 5 years. Thus, MCI represents a critical window of opportunity for intervening and altering the trajectory of both cognitive decline and loss of functional independence in older adults. Cognitive function apart from memory such as executive function is also impaired in patients with MCI. However, no study has yet placed sufficient emphasis on the training of executive function.

Objectives:

The objective of the study is to evaluate whether memory training combined with executive training could lead to improved cognitive and noncognitive performance in patients with MCI. Furthermore, we will explore the neural correlates underlying the changed performances.

Patients and Methods:

The proposed study is a single blinded, randomized and controlled trial that will include 120 elderly patients with MCI from the memory clinic. The groups will be randomized to either intervention or waiting-list group. The intervention is computerized combined memory and executive function training performed for 60 minutes x 4 times/week over 26 weeks. A neuropsychological assessment will be administered at baseline and week 4, 12 and 26 after the intervention. The structural and functional MRI, EEG and NIRS will be performed at baseline and week 26 after intervention for a sub-study on the effect of cognitive training on brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. An objective cognition impairment (a Montreal Cognitive Assessment (MoCA) score < 26)
2. Preserved general cognitive function( an mini-mental state examination (MMSE) score of > 24)
3. Clinical Dementia Rating (CDR) = 0.5
4. Hamilton Depression Scale (HAMD) score of < 12
5. Intact activities of daily living (ADL score of <=26)
6. Schooling education > = 5 years)
7. Not meeting the diagnosis of dementia (according to the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10) and the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) Probable Alzheimer's Criteria

Exclusion Criteria:

1. Serious visual or hearing impairment;
2. Hachinski Ischemia Scale (HIS) >= 4;
3. Subjects with Axis I disorders listed in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV), any other neurological disorders that could affect cognitive function;
4. currently on titration of medications with cognitive enhancers or antidepressants;
5. having any physical condition that could preclude regular attendance and full intervention-program participation

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite working memory z score | Change from baseline composite working memory z score at week 26
  composite score of digit span and spatial span

SECONDARY OUTCOMES:
cognitive test package (CTP) | Changes from baseline composite CTP score at week 26
  composite score of episodic memory, speed processing, executive function, attention, language and social cognition
Self evaluated memory ability | Change from baseline self evaluated memory ability at week 26
  Score on the questionnaire probes worries about memory (MMQ-contentment).
Brain Functional Imaging | change from baseline functional connectivity at week 26
  Brain function measured with MRI.
Electrical activity of the brain | change from baseline electrical brain activity at week 26
  Brain activity measured with electroencephalography (EEG).
Brain structural imaging | change from baseline cortical thickness at week 26
  cortical thickness measured with MRI
cerebral blood flow | change from baseline cerebral blood flow at week 26
  Cerebral blood flow measured with Near-infrared spectroscopy (NIRS).
Mood | Change from baseline composite mood score at week 26
  composite score of mood status
BDNF level | change from baseline serum BDNF level at week 26
  Serum Brain-derived neurotrophic factor (BDNF) level
Composite of overall cognition z scores | Changes from baseline composite overall cognition z score at week 26
  Score on Montreal Cognitive Assessment (MoCA) and Mini-mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Overall Officials: Huali Wang, MD, Principal Investigator — Peking University Institute of Mental Health(Sixth hospital)
Locations (1):
- Peking University Institute of Mental Health(Six Hospital), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Wang J, Sun T, Wang Z, Lyu X, Yu X, Wang H. A randomized controlled trial of combined executive function and memory training on the cognitive and noncognitive function of individuals with mild cognitive impairment: Study rationale and protocol design. Alzheimers Dement (N Y). 2018 Oct 15;4:556-564. doi: 10.1016/j.trci.2018.09.004. eCollection 2018. PMID 30386820